CLINICAL TRIAL: NCT00445705
Title: Safety and Efficacy of AGN 203818 for Pain Associated With Fibromyalgia Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated early due to company decision. Part B was never conducted.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 203818-503
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Results first posted 2012-01-20 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-08

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo (Placebo Comparator): Part A: Placebo every 12 hours for 4 weeks
  Interventions: Drug: placebo
- AGN 203818 3 mg (Experimental): Part A: 3 mg AGN 203818 every 12 hours for 4 weeks
  Interventions: Drug: AGN 203818
- AGN 203818 20 mg (Experimental): Part A: 20 mg AGN 203818 every 12 hours for 4 weeks
  Interventions: Drug: AGN 203818
- AGN 203818 60 mg (Experimental): Part A: 60 mg AGN 203818 every 12 hours for 4 weeks
  Interventions: Drug: AGN 203818

INTERVENTIONS:
Drug: placebo — Part A: Placebo every 12 hours for 4 weeks
  Arms: Placebo
Drug: AGN 203818 — Part A: AGN 203818 3 mg every 12 hours for 4 weeks
  Arms: AGN 203818 3 mg
Drug: AGN 203818 — Part A: AGN 203818 20 mg every 12 hours for 4 weeks
  Arms: AGN 203818 20 mg
Drug: AGN 203818 — Part A: AGN 203818 60 mg every 12 hours for 4 weeks
  Arms: AGN 203818 60 mg

SUMMARY:
This study will explore the safety and effectiveness of different doses of AGN 203818 in treating the pain associated with fibromyalgia syndrome. The study is being conducted in 2 parts. Part A enrolled 211 pts dosed with either 3, 20, 60 mg BID AGN 203818 or placebo over 4 week treatment duration. Part B will enroll 440 pts and dose with either 20, 100, 160 mg BID AGN 203818 or placebo over 12 week treatment duration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibromyalgia syndrome
* Moderate or severe pain associated with fibromyalgia

Exclusion Criteria:

* Any other uncontrolled disease
* Pregnant or nursing females

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2007-03; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (3):
- Canton, Ohio, United States
- Geneva, Switzerland
- Stanmore, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | AGN 203818 3 mg | AGN 203818 20 mg | AGN 203818 60 mg
Started | 53 | 53 | 52 | 53
Completed | 44 | 42 | 41 | 39
Not Completed | 9 | 11 | 11 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AGN 203818 3 mg | AGN 203818 20 mg | AGN 203818 60 mg | Total
Number analyzed (Participants) | 53 | 53 | 52 | 53 | 211
Age, Continuous [Median (Full Range); unit: years] | 50.5 [23 to 68] | 50.0 [25 to 69] | 49.5 [18 to 67] | 51.0 [24 to 71] | 50.0 [18 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 53 | 52 | 53 | 211
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Daily-Average-Pain Score at Week 4
Description: Change from Baseline in mean daily-average-pain score at week 4. Patients recorded their daily average pain on a 11-point scale (where 0 equals no pain and 10 equals worst pain imaginable) using a diary during the 4-week treatment period. A negative number change from baseline represents a decrease in average pain (improvement).
Time Frame: Baseline, Week 4
Population: Modified Intent-To-Treat (m-ITT). The m-ITT population included all patients who started the study (randomized) and received study medication with at least one post-treatment mean daily-average-pain score.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | AGN 203818 3 mg | AGN 203818 20 mg | AGN 203818 60 mg
Number analyzed (Participants) | 50 | 51 | 50 | 50
Scores on a Scale
  Baseline | 6.7 (1.04) | 6.7 (1.10) | 6.6 (0.96) | 6.7 (1.14)
  Change from Baseline at Week 4 | -1.3 (1.66) | -1.2 (1.82) | -1.5 (1.79) | -1.5 (1.85)

2. Secondary Outcome: Change From Baseline in the Short Form Brief Pain Inventory (SF-BPI) Average Pain Score at Week 4
Description: Change from baseline in the SF-BPI average pain question score at week 4. The SF-BPI is a patient-rated questionnaire that assesses certain aspects of pain including location, intensity, and interference with certain daily activities. The "average pain" question was rated on an 11-point scale (where 0=no pain and 10=worst pain imaginable). A negative number change from baseline indicates a reduction in average pain.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | AGN 203818 3 mg | AGN 203818 20 mg | AGN 203818 60 mg
Number analyzed (Participants) | 50 | 51 | 50 | 50
Scores on a Scale
  Baseline | 6.4 (1.19) | 6.6 (1.21) | 6.5 (1.23) | 6.5 (1.28)
  Change from Baseline at Week 4 | -1.3 (1.88) | -1.2 (1.79) | -1.7 (2.24) | -1.3 (1.68)

3. Secondary Outcome: Change From Baseline in the Fibromyalgia Impact Questionnaire (FIQ) Total Score of Physical Impairment at Week 4
Description: Change from baseline in FIQ total score of physical impairment at week 4. The FIQ is a disease-specific questionnaire consisting of 10 questions and visual analog scales regarding functional disability, pain intensity, sleep function, stiffness, anxiety, depression, and overall sense of wellbeing. Each question is scored from 0 to 10 with 0 = no impairment (best) and 10 indicates maximum impairment (worst), for a minimum possible score (best) of 0 and a maximum possible (worst) total score of 100. A negative number change from baseline indicates improvement.
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo | AGN 203818 3 mg | AGN 203818 20 mg | AGN 203818 60 mg
Number analyzed (Participants) | 50 | 51 | 50 | 50
Scores on a Scale
  Baseline | 59.9 (15.35) | 65.5 (15.55) | 65.7 (13.63) | 63.0 (13.44)
  Change from Baseline at Week 4 | -13.3 (16.67) | -15.1 (18.17) | -18.7 (20.51) | -12.8 (20.41)

4. Secondary Outcome: Patient Global Impression of Change (PGIC) for Fibromyalgia Syndrome Status at Week 4
Description: PGIC status for fibromyalgia syndrome at week 4. The PGIC consists of a self-evaluation by the patient of the overall change of their fibromyalgia syndrome since the beginning of the study, rated on a 7-point scale (score of 1-3 = very much improved to minimally improved; 4= no change; 5-7 = minimally worse to very much worse). Results are presented for the percentage of patients reporting each status: "improved"= score of 1-3; "no change"=score of 4; and "worse"=score of 5-7.
Time Frame: Week 4
Population: Modified Intent-To-Treat (m-ITT). The m-ITT population included all randomized patients who started study (randomized) and who received the study medication with at least one post-treatment mean daily-average-pain score.
Measure: Number; unit: Percentage of Patients
Arm/Group | Placebo | AGN 203818 3 mg | AGN 203818 20 mg | AGN 203818 60 mg
Number analyzed (Participants) | 50 | 51 | 50 | 50
Percentage of Patients
  Improved | 69.8 | 67.4 | 69.1 | 69.1
  No Change | 18.6 | 21.7 | 23.8 | 19.0
  Worse | 11.6 | 10.9 | 7.1 | 11.9

ADVERSE EVENTS:
Description: The safety population was used to calculate the number of participants at risk for SAEs and AEs and is the total number of patients that were randomized AND treated.
Arm/Group | Placebo | AGN 203818 3 mg | AGN 203818 20 mg | AGN 203818 60 mg
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/53 | 1/52 | 2/52
Other Adverse Events (participants affected / at risk) | 36/52 | 37/53 | 34/52 | 38/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=52) | AGN 203818 3 mg (N=53) | AGN 203818 20 mg (N=52) | AGN 203818 60 mg (N=52)
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=52) | AGN 203818 3 mg (N=53) | AGN 203818 20 mg (N=52) | AGN 203818 60 mg (N=52)
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 8
Nausea (Gastrointestinal disorders) | 5 | 8 | 7 | 5
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 0 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 1 | 0
Fatigue (General disorders) | 3 | 4 | 5 | 4
Oedema peripheral (General disorders) | 1 | 2 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 5 | 5 | 1 | 4
Nasopharyngitis (Infections and infestations) | 3 | 5 | 2 | 1
Urinary tract infection (Infections and infestations) | 3 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0
Headache (Nervous system disorders) | 7 | 13 | 9 | 13
Dizziness (Nervous system disorders) | 3 | 5 | 7 | 9
Somnolence (Nervous system disorders) | 1 | 4 | 4 | 6
Migraine (Nervous system disorders) | 3 | 3 | 0 | 0

LIMITATIONS AND CAVEATS:
This study was terminated early due to company decision. Only Part A results are presented; Part B was never conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo